CLINICAL TRIAL: NCT03658967
Title: Phase 2, Double-Blind, Placebo-Controlled, Randomized Efficacy, Safety and Tolerability Study of Lymfactin in Combination With Surgical Lymph Node Transfer To Patients With Secondary Lymphedema Associated With the Treatment of Breast Cancer
Brief Title: Clinical Study With Lymfactin® in the Treatment of Patients With Secondary Lymphedema (AdeLE)
Acronym: AdeLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herantis Pharma Plc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-LY-CL-2063; 2017-004443-20 (EudraCT Number)
Record Dates: First submitted 2018-07-06; First posted 2018-09-06 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Secondary Lymphedema
Keywords: Lymphedema; Breast cancer; Adenoviral vector; VEGF-C
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lymfactin® (1x10E11 vp) (Active Comparator): Lymfactin® will be administered as a single dose via perinodal injection in a volume of 2 mL.
  Interventions: Drug: Lymfactin® (1x10E11 vp)
- Placebo (0.9% physiological saline) (Placebo Comparator): Placebo will be administered as a single dose via perinodal injection in a volume of 2 mL.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lymfactin® (1x10E11 vp) — Lymfactin® will be administered as a single dose via perinodal injection in a volume of 2 mL.
  Other Names: LX-1101, AdAptVEGF-C adenoviral vector
  Arms: Lymfactin® (1x10E11 vp)
Drug: Placebo — Placebo will be administered as a single dose via perinodal injection in a volume of 2 mL.
  Other Names: 0.9% Physiological saline
  Arms: Placebo (0.9% physiological saline)

SUMMARY:
This study evaluates the efficacy of Lymfactin® in patients with secondary lymphedema associated with the treatment of breast cancer by comparing the effects of active study treatment Lymfactin® to placebo. The study product will be administered in combination with a surgical lymph node transfer operation. In addition, the safety and tolerability of the Lymfactin® treatment will be evaluated.

DETAILED DESCRIPTION:
This is a Phase II, double-blind, placebo-controlled, multi-centre clinical study, in which 40 patients with breast cancer associated secondary lymphedema will be randomized 1:1 either to Lymfactin® (1 x 10E11 viral particles, vp) or placebo (0.9% physiological saline) group.

The study product (Lymfactin® or placebo solution) will be administered as a single dose in a volume of two (2) mL, by ex vivo perinodal injection into the fat pad of a flap of tissue containing lymph nodes from the patient's own abdominal wall or the groin area. This flap of tissue will then be surgically implanted into the axillary region of the affected arm. This treatment with the study product is performed in combination with a surgical lymph node transfer, in conjunction with or without breast reconstruction surgery.

Patients will be followed-up for efficacy and safety according to a specified schedule up to 5 years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients with secondary lymphedema associated with the treatment of breast cancer and

   * Has undergone sentinel lymph node biopsies and/or lymph node resection in the axilla on the affected side of their breast cancer with initial N1-N2a staging and lymph node metastasis in ≤ 9 axillary lymph nodes.
   * Requires garment use as a compression treatment for the lymphedema in the affected arm.
   * Has the volume of the affected arm at least 10% greater than the unaffected arm following 7 days without compression garment.
   * Has the presence of pitting edema in the affected arm without compression garment.
   * Has had lymphedema for less than 5 years.
2. No evidence of recurrent or active breast cancer for at least 2 years after the breast cancer surgery and/or the end of chemotherapy and/or radiotherapy (excluding endocrine treatment).
3. Patient understands and voluntarily signs the written informed consent prior to any screening procedure.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
5. Body Mass Index (BMI) between 18 and 32 inclusive.
6. Positron Emission Tomography-Computed Tomography (PET CT) scan of the chest and the abdomen within 45 days before the study treatment without signs of active breast cancer or any other malignancy.
7. Adequate hematologic and end-organ function.

   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x the institutional upper limit of normal (ULN)
   * Bilirubin ≤ 1.5 x ULN (except in patients with previously documented Gilbert's syndrome, in which case total bilirubin ≤ 3 x ULN)
   * International Normalized ratio (INR) and Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 x ULN (for patients requiring therapeutic anticoagulation therapy, a stable INR ≤ 2,5)
   * Serum creatinine ≤ 1,5 x ULN or creatinine clearance ≥ 50 ml/min
   * Absolute neutrophil count (ANC) ≥ 1,5 E9/l
   * Platelet count ≥ 100 E9/l
   * Hemoglobin ≥ 100 g/l
8. Willingness to comply with scheduled visits, laboratory assessments, and other study-related procedures due to the regulatory requirements related to gene based therapies.
9. Non-smoker or willing to stop smoking or use of nicotine-containing products for at least 4 weeks prior to the study entry.
10. Negative urine pregnancy test (only patients with childbearing potential) at screening and use of adequate contraceptive measures from screening until six months after the study treatment administration:

    * A patient with childbearing potential should be using a reliable contraception method: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal, progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device (IUD), intrauterine hormone releasing system (IUS), bilateral tubal occlusion, vasectomised partner or sexual abstinence defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments.
    * A male patient is not allowed to donate sperm.
    * A patient with no current heterosexual relationship may be included according to the judgement of the Investigator.
    * For patient in postmenopausal state neither contraception nor a pregnancy test is required. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy.
    * For permanently sterile patient neither contraception nor a pregnancy test is required. A permanently sterile is defined by history of hysterectomy, bilateral salpingectomy or bilateral oophorectomy.

Exclusion Criteria:

1. Diagnosed for T4 and/or N2b/N3 stage breast cancer at the time of the original diagnosis.
2. Evidence (clinical, laboratory or imaging) or history of a neoplasm other than breast cancer (except basal cell carcinoma or cervical in situ carcinoma).
3. Diagnosed for metastatic breast cancer.
4. Pregnancy, lactation or a positive or indeterminate pregnancy test.
5. Current treatment with Cyclooxygenase-2 (COX-2) inhibitors should be interrupted from 2 weeks prior until 4 weeks post-treatment.
6. Previous treatment with, or participation in a trial of a gene therapy product.
7. Participation in a clinical trial, which has included interventions in the preceding 6 months or will involve future interventions. Participation in a non-interventional clinical trial, or in a non-interventional follow-up of any clinical trial, does not make the patient inappropriate for the entry into this study.
8. Current treatment with immunosuppressive drugs.
9. Current history of drug abuse, including nicotine-containing products, or alcohol abuse.
10. Known human immunodeficiency virus- or acquired immunodeficiency syndrome-related illness.
11. History of hepatic dysfunction, cirrhosis, or hepatitis.
12. Allergy to any ingredients of the Lymfactin® solution for injection.
13. Other concurrent severe acute and/or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with the study participation or study drug administration, that would, in the Investigator's judgement, affect the patient's ability to follow study-related procedures, or that may interfere with the interpretation of study results and would make the patient inappropriate for the entry into this study.
14. Doubtful availability, in the opinion of the Investigator, to complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Measurement of the volume of the arms | 24 Months
  Changes in the volume of the affected arm and comparison to the unaffected arm.
Measurement of the lymphatic flow of the affected arm by quantitative lymphoscintigraphy (99Tc-nanocolloid clearance rate with calculation of transport index). | 24 Months
  Assessment of the changes in the lymphatic flow.
Questionnaire according to the Lymphedema Quality of Life Inventory (LQOLI) | 24 Months
  Assessment of changes in the quality of life using Lymphedema Quality of Life Inventory (LQOLI) in which the patients assess how their lymphedema is affecting the activities of daily living. LQOLI consists of three dimensions: Physical, psychosocial and practical, which are reported separately as the mean score of that part. Each part of the LQOLI is scored from 0 to 3, where score 0 means "no impact", 1 means "a little bit impact", 2 means "somewhat impact" and score 3 means "significant impact" on the quality of life of the patient, the smaller score thus being the better.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 Months
  Adverse Events as assessed by CTCAE v4.0 to evaluate the safety profile after administration of Lymfactin.
CT scan of chest and abdomen | 60 Months
  Changes in CT scans of chest and abdomen in order to detect malignancies.
Lymfactin genome copy number in blood | 30 Days
  Changes in Lymfactin genome copy number in blood.
Lymfactin genome copy number in wound secretion | 7 Days
  Changes in Lymfactin genome copy number in wound secretion.
Formation of anti-Lymfactin antibodies | 12 Months
  Changes in anti-Lymfactin antibody titer in blood.
Systemic concentration of vascular endothelial growth factor C (VEGF-C) | 30 Days
  Changes in the VEGF-C concentration in blood.

OTHER OUTCOMES:
Optional evaluation of the anatomy and functionality of lymphatic vessels by MRI lymphangiography | 24 Months
  Changes in anatomy and functionality of lymphatic vessels by newly developed MRI lymphangiography and comparison of the correlation of the method to the already established lymphoscintigraphy in the assessment of lymphedema.
Percentage Water Content (PWC) measurement of water content and edema | 24 months
  Changes in PWC measurement of water content and edema in affected arm and comparison to the unaffected arm.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Saarikko, MD, PhD, Principal Investigator — Helsinki University Central Hospital; Maria Mani, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (5):
- Finland (3):
  - Töölö Hospital, Department of Plastic Surgery, Helsinki
  - Tampere University Hospital, Department of Plastic Surgery, Tampere
  - Turku University Hospital, Department of Plastic Surgery, Turku
- Sweden (2):
  - Karolinska University Hospital, Department of Reconstructive Plastic Surgery, Stockholm
  - Uppsala University Hospital, Department of Plastic Surgery, Uppsala